CLINICAL TRIAL: NCT06523478
Title: A Study on the Efficacy and Safety of Intratonsillar Immunotherapy for Allergic Rhinitis
Brief Title: Intratonsillar Immunotherapy for Allergic Rhinitis
Acronym: ITITFAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xu Yu (Other)
Responsible Party: Sponsor-Investigator, Xu Yu, Professor, Chief Physician, Renmin Hospital of Wuhan University
Organization: Renmin Hospital of Wuhan University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WDRY2024-K097; 2021-1-X-2 (Other: Wuhan University Renmin Hospital)
Record Dates: First submitted 2024-07-18; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Allergic Rhinitis
Keywords: Allergic rhinitis; Intratonsillar; Allergen immunotherapy; Standardized dust mite allergen extracts
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Masking Description: This experiment is a comparative study of two treatment methods, and there are obvious differences between the treatment methods of the experimental group and the control group, so it is difficult to blind the subjects, researchers and evaluators, and only the experiment design without blindness can be adopted.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intratonsillar Immunotherapy (ITIT) group (Experimental): The intervention of ITIT will be a series of 3 injections of a commercially-available standardized dust mite allergen extracts (Novo Helisen-Depot, Allergopharma, Merck, Germany) given every four weeks into tonsil through guidance using a 1-mL hypodermic syringe with a 25-gauge or smaller needle. The specific doses are 5 TU (0.1 ml, the first injection), 50 TU (0.1 ml, the second injection), and 50 TU (0.1 ml, the third injection).
  Before each injection, patients will take one tablet of antihistamine.
  Interventions: Procedure: Intratonsillar immunotherapy (ITIT)
- Subcutaneous Immunotherapy (SCIT) group (Active Comparator): The same drugs will be used in active comparator. SCIT consists of two stages: the accumulation stage and the maintenance stage. During the initial 14 weeks, patients will receive sequential subcutaneous injections as follows: (1) 1st vial: 0.1 mL, 0.2 mL, 0.4 mL, and 0.8 mL; (2) 2nd vial: 0.1 mL, 0.2 mL, 0.4 mL, and 0.8 mL; (3) 3rd vial: 0.1 mL, 0.2 mL, 0.4 mL, 0.6 mL, 0.8 mL, and 1.0 mL of allergen, achieving a maintenance dose of 5000 TU. Subsequently, maintenance therapy involves subcutaneous injections of 5000 TU (1.0 mL, 3rd vial) every 4-6 weeks. The intervention process before and after each injection is similar to that of the ITIT group.
  Interventions: Procedure: Subcutaneous immunotherapy (SCIT)

INTERVENTIONS:
Procedure: Intratonsillar immunotherapy (ITIT) — During injection, the operator needs to gently shake the injection bottle about 20 times, the drug must be mixed to ensure the consistency of allergen concentration, and carefully check the patient's name and concentration on the bottle. Allergy extracts should not be injected intravenously, so the syringe will be aspirated to avoid inadvertent intravascular injection. Before each injection, after inserting the needle into the selected tonsil, before injecting the dose, the investigator will slightly pull the plunger of the syringe. If blood returns from the syringe, the syringe, and its contents will be discarded. The other tonsil will be selected and a new syringe will be prepared.
  Arms: Intratonsillar Immunotherapy (ITIT) group
Procedure: Subcutaneous immunotherapy (SCIT) — Injection requires shaking bottle 20x to mix drug for consistency. Verify patient name & concentration. Use 1 ml skin test syringe for deep subcutaneous injection at 45° angle, 1 cm into outer upper arm. Lift skin folds for deeper injection, avoid subcutaneous, muscular or intravascular. Inject slowly, 1 min for 1 ml. Avoid shallow injections which may cause local side effects. Alternate between left & right arm for 5 min after injection for compression.
  Arms: Subcutaneous Immunotherapy (SCIT) group

SUMMARY:
This is a prospective, open-label, positive parallel controlled, blinded endpoint clinical study designed to compare the safety and efficacy of "Intratonsillar Immunotherapy of Standardized Dust Mite Allergen Extracts (Novo Helisen-Depot, Allergopharma, Merck, Germany)" with Subcutaneous Immunotherapy in patients with "Dust Mite Allergic Rhinitis."

Participants will be evaluated for safety and efficacy throughout the entire three-year period.

DETAILED DESCRIPTION:
Background:

Allergic Rhinitis (AR) presents both nasal and non-nasal symptoms. The global incidence of AR is rising, causing a significant burden. Seasonal allergic rhinitis (SAR) and perennial allergic rhinitis (PAR) are the two related clinical divisions of AR. Allergen immunotherapy (AIT) is a treatment involving the injection of specific allergens into the body. Studies have evaluated the effectiveness and safety of subcutaneous (SCIT), sublingual (SLIT), and intra-lymphatic immunotherapy (ILIT). The mechanisms underlying AIT involve both innate and acquired immunity. AIT modulates the activity of various immune cells, including dendritic cells, innate lymphoid cells (ILCs), and regulatory T cells (Tregs).

Intra-lymphatic inoculation (ILIT) has been studied in animals for its ability to improve T cell response to antigens. Studies have found that direct injection of antigens into lymph nodes can lead to improved T cell response and more efficient delivery of the antigen to subcutaneous lymph nodes. ILIT has been effective in treating atopic dermatitis, producing targeted IgG antibodies, enhancing lymphocyte responses, and treating viral and tumor challenges. It has also been effective in treating allergies and reducing symptoms of allergic rhinitis in mice. Studies have found ILIT to be effective in treating atopic dermatitis in dogs caused by common allergens and insect bite hypersensitivity in horses caused by biting midges. In general, animal studies support the use of ILIT as a safe and effective means to induce IgG and T cell responses with fewer treatments and lower doses compared to subcutaneous injection across a range of species.

Objectives:

The primary objective is to explore the efficacy, clinical value, and possible mechanism of action of Intratonsillar Immunotherapy (ITIT) by recording and analyzing the questionnaire scores after ITIT versus SCIT, while comparing the trend of bio-indicator changes in these two treatments.

Primary Endpoint:

Combined Symptom and Medication Score (CSMS): CSMS serves as the primary efficacy endpoint, tracking changes in participant symptoms and assessing the sustainability and stability of treatment effects. It comprises:

Allergen-induced symptom score: Scored from 0 (no symptoms) to 3 (most severe symptoms) for nasal congestion, rhinorrhea, nasal itching, sneezing, eye itching, and tearing, with the average yielding the symptom score (SS).

Emergency medication use related to allergy symptoms: Assigned points based on antihistamine (1 point/day), nasal corticosteroid (2 points/day), and oral corticosteroid (3 points/day) usage, with the highest value determining the medication score (MS).

CSMS (0-6) = SS (0-3) + MS (0-3). Recorded at baseline and 1, 2, 3, 6, 12, 24, and 36 months post-dust mite extract treatment.

Adverse Reactions: Participants were observed for 30 minutes post-injection and encouraged to report any adverse events during follow-up. Adverse reactions were classified as local (LR) or systemic (SR) according to the World Allergy Organization Subcutaneous Immunotherapy Response Classification System. Detailed records included occurrence time, number of injections, clinical manifestations, and management measures.

Study Population:

A total of 120 screened participants will be required to enroll 60 subjects in each group, with an age range of 5-65 years.

Sites/Facilities Enrolling Participants:

Renmin Hospital of Wuhan University will recruit participants.

Description of Study Intervention:

In this study, participants who meet the enrollment criteria will be randomly assigned to two groups. The random assignment will be performed by an independent investigator using a computer-generated sequence of random numbers. The assignment process will be conducted before participants are enrolled to ensure fairness and randomness in the grouping. Each group will be assigned an equal number of participants to ensure the objectivity and comparability of the studies.

Due to the obvious differences between the treatment methods of the experimental group and the control group, it is difficult to blind the subjects, researchers, and evaluators. Therefore, a non-blind experimental design is adopted. To minimize bias, blind data review will be employed.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily sign informed consent.
* Commitment to follow the research procedures and cooperate with the implementation of the entire research process.
* Diagnosis in accordance with ARIA guidelines, based on:

  ① Symptoms: Two or more symptoms such as paroxysmal sneezing, watery nose, nasal itching, and nasal congestion, with symptoms lasting or accumulating for more than 1 hour per day. May be accompanied by eye symptoms such as tearing, eye itching, and eye redness.

  ② Signs: Common nasal mucosa pale, edema, nasal watery secretions.
  * Allergen test: Positive for skin prick test (SPT) and/or serum-specific IgE for at least one allergen, or positive for nasal provocation test.
* Have a history of allergic rhinitis caused by atopic allergens and one of the following:

  ① No significant relief after drug treatment.

  ② Do not want to continue taking medication for a long time.

  ③ Long-term drug treatment can produce adverse side effects.
  * Allergens cannot be effectively avoided in daily life.
* Women of childbearing age must ensure that they do not become pregnant during the treatment cycle.
* Must be between 5 and 65 years old.

Exclusion Criteria:

* Allergic to the excipient (aluminum hydroxide) of Allergopharma or the rescue medication epinephrine.
* Respiratory disease other than stable asthma.
* Pulmonary insufficiency (NYHA grade II and above or FEV1 < 80%) or irreversible changes in the responding organs such as emphysema and bronchiectasis.
* Severe acute or chronic diseases (including malignant diseases), inflammation, and fever.
* Multiple sclerosis.
* Immune system diseases (autoimmune diseases, immune diseases caused by antigen and antibody complexes, immune deficiencies, etc.).
* Active tuberculosis.
* Severe mental disorder.
* Obvious cardiac insufficiency.
* A history of severe recurrent acute sinusitis (defined as two episodes per year within the past 2 years, each requiring antibiotic treatment).
* A history of chronic sinusitis, including at least two of the following symptoms (at least one of which should be nasal congestion or runny nose):

  ① Nasal congestion, runny nose, facial pressure, or pain.

  ② Having a diminished or lost sense of smell.

  ③ Endoscopic or CT examination showed signs of sinusitis.
* Severe liver and renal impairment, including but not limited to abnormal liver function (such as ALT, AST elevation more than 2 times the normal range), abnormal kidney function (such as creatinine clearance less than 60 mL/min), etc.
* Smokers averaging more than 5 cigarettes per day in the 3 months prior to the trial or unable to give up smoking during the entire hospital stay.
* Regular drinkers in the 3 months prior to the trial, i.e., more than 2 units of alcohol per day on average (1 unit = 360ml beer or 45ml spirits with 40% alcohol or 150ml wine).
* Received immunotherapy within the last 3 years (subcutaneous injection or sublingual allergen-specific immunotherapy, etc.).
* Patients who used experimental drugs or participated in other clinical studies within 30 days prior to treatment.
* Patients treated with IgE monoclonal antibodies within the last 4 months.
* Patients who are taking beta blockers.
* Patients who do not have sufficient knowledge about the trial.
* Not between the ages of 5 and 65.
* Patients who are pregnant or nursing during the study period, or who plan to become pregnant.
* Patients who are unable to have tonsil injections due to chronic tonsillitis, small tonsils, prior tonsillectomy, etc.

Ages: 5 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-04-29 (Actual); Primary Completion 2028-04-29 (Estimated); Study Completion 2028-04-29 (Estimated)

PRIMARY OUTCOMES:
Combined Symptom and Medication Score (CSMS) | Pre-intervention screening period; 3 months, 6 months, 12 months, 24 months, 36 months after the first intervention. Up to 36 months
  Combined Symptom and Medication Score (CSMS) serves as the primary efficacy endpoint, tracking changes in participant symptoms and assessing the sustainability and stability of treatment effects. It comprises:
  Allergen-induced symptom score: Scored from 0 (no symptoms) to 3 (most severe symptoms) for nasal congestion, rhinorrhea, nasal itching, sneezing, eye itching, and tearing, with the average yielding the symptom score (SS).
  Emergency medication use related to allergy symptoms: Assigned points based on antihistamine (1 point/day), nasal corticosteroid (2 points/day), and oral corticosteroid (3 points/day) usage, with the highest value determining the medication score (MS).
  CSMS (0-6) = SS (0-3) + MS (0-3). Recorded at baseline and 1, 2, 3, 6, 12, 24, and 36 months post-dust mite extract treatment.
Number of Participants with Local or Systemic Adverse Reactions | After each treatment. Up to 36 months
  Participants will be observed for 30 minutes post-injection and encouraged to report any adverse events during follow-up. Adverse reactions are classified as local reaction (LR) or systemic reaction (SR) according to the World Allergy Organization Subcutaneous Immunotherapy Response Classification System. Detailed records include occurrence time, number of injections, clinical manifestations, and management measures.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | Pre-intervention screening period; 3 months, 6 months, 12 months, 24 months, 36 months after the first intervention. Up to 36 months
  Pain perception of allergy symptoms during treatment will be evaluated using a scale ranging from 0 to 10, where 0 indicates no pain and 10 indicates maximum pain.
Absolute Value and Percentage of Blood Leukocytes | Pre-intervention screening period; 3 months, 6 months, 12 months, 24 months, 36 months after the first intervention. Up to 36 months
  Changes in blood eosinophil absolute value (EOS), eosinophil percentage (EOS%), basophil absolute value (BAS), and basophil percentage (BAS%) will be evaluated.
Concentration of Key Serum Cytokines | Pre-intervention screening period; 3 months, 6 months, 12 months, 24 months, 36 months after the first intervention. Up to 36 months
  Changes in key serum cytokines, including TNF-α, IFN-γ, IL-2, IL-4, IL-6, IL-10, and IL-17, will be evaluated at the same intervals as CSMS.
Concentration of Serum Immune Globulins | Pre-intervention screening period; 3 months, 6 months, 12 months, 24 months, 36 months after the first intervention. Up to 36 months
  Changes in serum total IgE (tIgE), IgA, IgG, and specific IgE (sIgE) will be evaluated at the same intervals as CSMS.
Proportion of Blood T Cell Differentiation | Pre-intervention screening period; 3 months, 6 months, 12 months, 24 months, 36 months after the first intervention. Up to 36 months
  Changes in the proportion of blood T cell differentiation (Th, Tfh, Tfr, Treg, Tfc, Tex, etc.) will be evaluated.
RQLQ | Pre-intervention screening period; 3 months, 6 months, 12 months, 24 months, 36 months after the first intervention. Up to 36 months
  Administration of questionnaires, the Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ).
Concentration of FeNO | Pre-intervention screening period; 3 months, 6 months, 12 months, 24 months, 36 months after the first intervention. Up to 36 months
  Change of FeNO

CONTACTS AND LOCATIONS:
Overall Officials: Yu Xu, Study Chair — Renmin Hospital of Wuhan University
Locations (1):
- Renmin Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
Two years after the completion of the trial, data will be published on the EDC of Metz Medical (https://edc-cloud.medsci.cn/).
Supporting Information: Study Protocol, CSR
Time Frame: Two years after the completion of the trial
Access Criteria: Upon approval of the request, access to the de-identified individual patient-level data will be provided. Before accessing the requested information, a data sharing agreement (a non-negotiable contract for data visitors) must be signed.
URL: http://edc-cloud.medsci.cn/

REFERENCES:
- [Background] Waage J, Standl M, Curtin JA, Jessen LE, Thorsen J, Tian C, Schoettler N; 23andMe Research Team; AAGC collaborators; Flores C, Abdellaoui A, Ahluwalia TS, Alves AC, Amaral AFS, Anto JM, Arnold A, Barreto-Luis A, Baurecht H, van Beijsterveldt CEM, Bleecker ER, Bonas-Guarch S, Boomsma DI, Brix S, Bunyavanich S, Burchard EG, Chen Z, Curjuric I, Custovic A, den Dekker HT, Dharmage SC, Dmitrieva J, Duijts L, Ege MJ, Gauderman WJ, Georges M, Gieger C, Gilliland F, Granell R, Gui H, Hansen T, Heinrich J, Henderson J, Hernandez-Pacheco N, Holt P, Imboden M, Jaddoe VWV, Jarvelin MR, Jarvis DL, Jensen KK, Jonsdottir I, Kabesch M, Kaprio J, Kumar A, Lee YA, Levin AM, Li X, Lorenzo-Diaz F, Melen E, Mercader JM, Meyers DA, Myers R, Nicolae DL, Nohr EA, Palviainen T, Paternoster L, Pennell CE, Pershagen G, Pino-Yanes M, Probst-Hensch NM, Ruschendorf F, Simpson A, Stefansson K, Sunyer J, Sveinbjornsson G, Thiering E, Thompson PJ, Torrent M, Torrents D, Tung JY, Wang CA, Weidinger S, Weiss S, Willemsen G, Williams LK, Ober C, Hinds DA, Ferreira MA, Bisgaard H, Strachan DP, Bonnelykke K. Genome-wide association and HLA fine-mapping studies identify risk loci and genetic pathways underlying allergic rhinitis. Nat Genet. 2018 Aug;50(8):1072-1080. doi: 10.1038/s41588-018-0157-1. Epub 2018 Jul 16. PMID 30013184
- [Background] Skoner DP. Allergic rhinitis: definition, epidemiology, pathophysiology, detection, and diagnosis. J Allergy Clin Immunol. 2001 Jul;108(1 Suppl):S2-8. doi: 10.1067/mai.2001.115569. PMID 11449200
- [Background] Smith JM, Pizarro YA. Hyposensitization with extracts of Dermatophagoides pteronyssinus and house dust. Clin Allergy. 1972 Sep;2(3):281-3. doi: 10.1111/j.1365-2222.1972.tb01291.x. No abstract available. PMID 4643787
- [Background] James C, Bernstein DI. Allergen immunotherapy: an updated review of safety. Curr Opin Allergy Clin Immunol. 2017 Feb;17(1):55-59. doi: 10.1097/ACI.0000000000000335. PMID 27906697
- [Background] Senti G, Prinz Vavricka BM, Erdmann I, Diaz MI, Markus R, McCormack SJ, Simard JJ, Wuthrich B, Crameri R, Graf N, Johansen P, Kundig TM. Intralymphatic allergen administration renders specific immunotherapy faster and safer: a randomized controlled trial. Proc Natl Acad Sci U S A. 2008 Nov 18;105(46):17908-12. doi: 10.1073/pnas.0803725105. Epub 2008 Nov 10. PMID 19001265
- [Background] Zimmer A, Bouley J, Le Mignon M, Pliquet E, Horiot S, Turfkruyer M, Baron-Bodo V, Horak F, Nony E, Louise A, Moussu H, Mascarell L, Moingeon P. A regulatory dendritic cell signature correlates with the clinical efficacy of allergen-specific sublingual immunotherapy. J Allergy Clin Immunol. 2012 Apr;129(4):1020-30. doi: 10.1016/j.jaci.2012.02.014. PMID 22464673
- [Background] Swamy RS, Reshamwala N, Hunter T, Vissamsetti S, Santos CB, Baroody FM, Hwang PH, Hoyte EG, Garcia MA, Nadeau KC. Epigenetic modifications and improved regulatory T-cell function in subjects undergoing dual sublingual immunotherapy. J Allergy Clin Immunol. 2012 Jul;130(1):215-24.e7. doi: 10.1016/j.jaci.2012.04.021. Epub 2012 Jun 5. PMID 22677046
- [Background] Rosskopf S, Jahn-Schmid B, Schmetterer KG, Zlabinger GJ, Steinberger P. PD-1 has a unique capacity to inhibit allergen-specific human CD4+ T cell responses. Sci Rep. 2018 Sep 10;8(1):13543. doi: 10.1038/s41598-018-31757-z. PMID 30201974
- [Background] Shamji MH, Larson D, Eifan A, Scadding GW, Qin T, Lawson K, Sever ML, Macfarlane E, Layhadi JA, Wurtzen PA, Parkin RV, Sanda S, Harris KM, Nepom GT, Togias A, Durham SR. Differential induction of allergen-specific IgA responses following timothy grass subcutaneous and sublingual immunotherapy. J Allergy Clin Immunol. 2021 Oct;148(4):1061-1071.e11. doi: 10.1016/j.jaci.2021.03.030. Epub 2021 Apr 2. PMID 33819508
- [Background] JUILLARD G, BUBBERS J E. Experimental intra-lymphatic immunotherapy (ILI) of canine allergic disease[C/OL]. 1983[2023-02-12]. https://www.semanticscholar.org/paper/Experimental-intra-lymphatic-immunotherapy-(ILI)-of-Juillard-Bubbers/3d454bcc0cb13e5375ac58a9f415672a0c6b609c.
- [Background] Sigel MB, Sinha YN, VanderLaan WP. Production of antibodies by inoculation into lymph nodes. Methods Enzymol. 1983;93:3-12. doi: 10.1016/s0076-6879(83)93031-8. PMID 6346012
- [Background] Maloy KJ, Erdmann I, Basch V, Sierro S, Kramps TA, Zinkernagel RM, Oehen S, Kundig TM. Intralymphatic immunization enhances DNA vaccination. Proc Natl Acad Sci U S A. 2001 Mar 13;98(6):3299-303. doi: 10.1073/pnas.051630798. Epub 2001 Feb 27. PMID 11248073
- [Background] Johansen P, Haffner AC, Koch F, Zepter K, Erdmann I, Maloy K, Simard JJ, Storni T, Senti G, Bot A, Wuthrich B, Kundig TM. Direct intralymphatic injection of peptide vaccines enhances immunogenicity. Eur J Immunol. 2005 Feb;35(2):568-74. doi: 10.1002/eji.200425599. PMID 15682446
- [Background] Martinez-Gomez JM, Johansen P, Erdmann I, Senti G, Crameri R, Kundig TM. Intralymphatic injections as a new administration route for allergen-specific immunotherapy. Int Arch Allergy Immunol. 2009;150(1):59-65. doi: 10.1159/000210381. Epub 2009 Apr 2. PMID 19339803
- [Background] Kreiter S, Selmi A, Diken M, Koslowski M, Britten CM, Huber C, Tureci O, Sahin U. Intranodal vaccination with naked antigen-encoding RNA elicits potent prophylactic and therapeutic antitumoral immunity. Cancer Res. 2010 Nov 15;70(22):9031-40. doi: 10.1158/0008-5472.CAN-10-0699. Epub 2010 Nov 2. PMID 21045153
- [Background] Kim EH, Kim JH, Samivel R, Bae JS, Chung YJ, Chung PS, Lee SE, Mo JH. Intralymphatic treatment of flagellin-ovalbumin mixture reduced allergic inflammation in murine model of allergic rhinitis. Allergy. 2016 May;71(5):629-39. doi: 10.1111/all.12839. Epub 2016 Feb 12. PMID 26752101
- [Background] Fischer N, Rostaher A, Favrot C. [Intralymphatic immunotherapy: An effective and safe alternative route for canine atopic dermatitis]. Schweiz Arch Tierheilkd. 2016 Sep;158(9):646-652. doi: 10.17236/sat00085. German. PMID 27655164
- [Background] Landolt GA, Hussey SB, Kreutzer K, Quintana A, Lunn DP. Low-dose DNA vaccination into the submandibular lymph nodes in ponies. Vet Rec. 2010 Aug 21;167(8):302-3. doi: 10.1136/vr.c3891. No abstract available. PMID 20729518
- [Background] Juillard GJ, Boyer PJ, Yamashiro CH. A phase I study of active specific intralymphatic immunotherapy (ASILI). Cancer. 1978 Jun;41(6):2215-25. doi: 10.1002/1097-0142(197806)41:63.0.co;2-x. PMID 77718
- [Background] Draube A, Klein-Gonzalez N, Mattheus S, Brillant C, Hellmich M, Engert A, von Bergwelt-Baildon M. Dendritic cell based tumor vaccination in prostate and renal cell cancer: a systematic review and meta-analysis. PLoS One. 2011 Apr 20;6(4):e18801. doi: 10.1371/journal.pone.0018801. PMID 21533099
- [Background] Schmid JM, Nezam H, Madsen HH, Schmitz A, Hoffmann HJ. Intralymphatic immunotherapy induces allergen specific plasmablasts and increases tolerance to skin prick testing in a pilot study. Clin Transl Allergy. 2016 May 25;6:19. doi: 10.1186/s13601-016-0107-x. eCollection 2016. PMID 27231527
- [Background] Patterson AM, Bonny AE, Shiels WE 2nd, Erwin EA. Three-injection intralymphatic immunotherapy in adolescents and young adults with grass pollen rhinoconjunctivitis. Ann Allergy Asthma Immunol. 2016 Feb;116(2):168-70. doi: 10.1016/j.anai.2015.11.010. Epub 2015 Dec 17. No abstract available. PMID 26706294
- [Background] Lee SP, Choi SJ, Joe E, Lee SM, Lee MW, Shim JW, Kim YJ, Kyung SY, Park JW, Jeong SH, Jung JH. A Pilot Study of Intralymphatic Immunotherapy for House Dust Mite, Cat, and Dog Allergies. Allergy Asthma Immunol Res. 2017 May;9(3):272-277. doi: 10.4168/aair.2017.9.3.272. PMID 28293934